CLINICAL TRIAL: NCT03778814
Title: TCR-T Cells Targeting Cancer Cells for Immunotherapy of Lung Cancer and Other Solid Tumors: Phase I Clinical Trial
Brief Title: TCR-T Cell Immunotherapy of Lung Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Tcell Immune (Guangzhou) Science and Technology Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZTCRT-006
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nonsmall Cell Lung Cancer; Solid Tumor, Adult
Keywords: Lung Cancer; Solid Tumor; Immunotherapy; TCR-T Cell Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cell therapy group (Experimental): Appropriate lung cancer or other solid tumor patients who could benefit from immunotherapy will be treated with targeting TCR-T cells.
  Interventions: Biological: TCR-T cells

INTERVENTIONS:
Biological: TCR-T cells — Engineering TCR-T cells targeting lung tumor and other solid tumor will be transfused back the patients.

SUMMARY:
Tumor organoids and TILs (and/or peripheral T cells) cultures will be established from fresh tissure of lung cancer and other solid tumors. Coculture will be utilized to screen tumor-responsive T cells which are further selected for monoclonal expansion and TCR cloning for engineered reconstitution of TCR-T cells. After verification by multiple in vitro and in vivo studies, a large number of TCR-T cells will be introduced back into the patients via vein, artery or fine needle punctured to the tumor, or combinations. In this phase I study, the safety, tolerance and preliminary efficacy of the TCR-T cell immunotherapy on human will firstly be assessed.

DETAILED DESCRIPTION:
1. Choose appropriate patients with KK-LC-1 expression in advanced lung cancer or other solid tumors and matched MHC-A11 typing, with written consent for this study; For cancer without expression of KK-LC-1, fresh tumor tissue should be obtained for RNA/DNA sequencing to computationally identify neoantigen peptides that can be captured by specifically personizedly synthesized poly-MHCI which can be further used to fish appropriate T cells from the patient.
2. Perform biopsy to obtain tissue from tumor/lymph node for organoids, TILs, DC and T cells culture, coculture to screening anti-tumor T cells, establish and select monoclonal T cells for TCR cloning;
3. Clone TCR sequence that targets KK-LC-1 or neoantigens; collect PBMCs from the blood of the patients, isolate and activate the T cells and generate the TCR-T cells;
4. Test the quality and killing activity of the TCR-T cells in vitro and then transplant back the patients via systemic (vein and/or artery) or local injections, and follow up closely to collect related clinical data as needed;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. patients with advanced lung tumor or other solid tumor where biopsy is obtainable
2. Life expectancy >12 weeks
3. Child-Pugh-Turcotte score <7
4. Adequate heart,lung,liver,kidney function
5. Available autologous transduced T cells with greater than or equal to 20% expression of targeted TCR sequences determined by flow-cytometry and killing of tumor cells greater than or equal to 20% in cytotoxicity assay
6. Informed consent explained to, understood by and signed by patient/ guardian. Patient/guardian given copy of informed consent. -

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Tumor size more than 25cm;
3. Severe virus infection such as HBV, HCV, HIV, et al
4. Known HIV positivity
5. History of lung transplantation
6. Active infectious disease related to bacteria, virus,fungi,et al
7. Other severe diseases that the investigators consider not appropriate;
8. Pregnant or lactating women
9. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
10. Other conditions that the investigators consider not appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2036-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | three months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the TCR-T cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission | three months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.

OTHER OUTCOMES:
Median TCR-T cell persistence | Five years
  Median TCR-T cell persistence will be measured by quantitative rt-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China